CLINICAL TRIAL: NCT06320886
Title: Role of Ultrasonography in Acute Abdomen in Adults in Correlation to Computed Tomography Scan
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Abdelmotalib, Radiologist, Sohag University
Other Study IDs: Soh-Med-24-02-05MS
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Acute Abdomen; In Adults
MeSH Terms: conditions — Abdomen, Acute | interventions — Diagnostic Tests, Routine; Ultrasonography; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic Test — Use both ultrasonography and Computed tomography scan to diagnose the causes of Acute Abdominal Pain in Adults.
  Other Names: ultrasonography and Computed Tomography Scan

SUMMARY:
The study aims to evaluate the role of Ultrasonography in the diagnosis of the cause of acute abdominal pain in 50 adults presenting in the ER at Sohag University Hospital and compares it to the Computed Tomography scan results of the same patients to discover the superiority of both over the other in the diagnosis of different acute abdomen cases.

ELIGIBILITY:
Inclusion Criteria:

* Adults presented with Acute abdominal pain.

Exclusion Criteria:

* less than 18 years old patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults presented to the ER of Sohag University Hospital with Acute abdominal pain, both Ultrasonography and Computed tomography are used to diagnose the causes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Comparison between the role of Ultrasonography and Computed Tomography in Acute Abdomen diagnosis | 6-9 Months
  evaluate the accuracy of both Ultrasonography and Computed Tomography Scan in diagnosis of Acute abdomen in adults

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt